CLINICAL TRIAL: NCT03685214
Title: Comparison of Balanced Crystalloids and Normal Saline in Septic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ZhiYong Peng (Other)
Collaborators: Wu Jieping Medical Foundation (Other)
Responsible Party: Sponsor-Investigator, ZhiYong Peng, Professor, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018010
Record Dates: First submitted 2018-08-15; First posted 2018-09-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2018-10

CONDITIONS: Sepsis; Acute Kidney Injury; Septic Shock; Sepsis, Severe
Keywords: sepsis; intensive care unit; acetated Ringer's solution; AKI; normal saline; prognosis; continuous renal replacement therapy
MeSH Terms: conditions — Sepsis; Acute Kidney Injury; Shock, Septic | interventions — Saline Solution; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: One model using normal saline for resuscitation fluid,the other using acetated Ringer's solution
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.9% saline (Experimental): We use 0.9% saline for resuscitation fluid in ICU septic patients
  Interventions: Drug: 0.9% saline
- Balanced Crystalloids (Experimental): We use acetated Ringer's solution for resuscitation fluid in ICU septic patients
  Interventions: Drug: lactated Ringer's solution

INTERVENTIONS:
Drug: 0.9% saline — we use 0.9% saline in ICU patients with sepsis for resuscitation fluid.
  Other Names: normal saline
  Arms: 0.9% saline
Drug: lactated Ringer's solution — we use balanced balanced crystalloids in ICU patients with sepsis for resuscitation fluid.
  Other Names: Ringer's lactate
  Arms: Balanced Crystalloids

SUMMARY:
In this prospective randomized controlled trial, investigators attempt to study the effects of acetated Ringer's solution on the prognosis and renal function of patients with sepsis in intensive care unit compared with normal saline, and provide evidence for current fluid resuscitation strategies for sepsis.

DETAILED DESCRIPTION:
During the study period，either normal saline or acetated Ringer's solution will be assigned as resuscitation fluid to the septic patients meeting the inclusion criteria.It is anticipated that about 500 patients will be enrolled during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed sepsis aged 18~75 and accepted therapy in ICU

Exclusion Criteria:

* Need of Renal replacement treatment
* End-stage renal failure
* pregnant woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Development of kidney injury as defined by the KDIGO criteria. | 5 days after the admission
  Investigators will use the level of creatinine(μmol/L) and body weight adjusted urine(ml/h/kg) for severity assessment of kidney injury
Need of renal replacement treatment | After the admission and before the discharge from ICU,average 15 days
  Investigators will assess patients' kidney function everyday

SECONDARY OUTCOMES:
ICU stay | After the admission and before the discharge from ICU,average 15 days
  the time of patients' requirement for critical care
28 days mortality | 28 days after the admission in ICU
  the short time mortality

CONTACTS AND LOCATIONS:
Overall Officials: ZhiYong Peng, professor, Study Director — Zhongnan Hospital
Locations (1):
- Zhongnan Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zhang J, Liu F, Wu Z, Jiang J, Wang B, Qian Y, Suo J, Li Y, Peng Z. ACETATE RINGER'S SOLUTION VERSUS NORMAL SALINE SOLUTION IN SEPSIS: A RANDOMIZED, CONTROLLED TRIAL. Shock. 2024 Apr 1;61(4):520-526. doi: 10.1097/SHK.0000000000002324. Epub 2024 Feb 1. PMID 38369528
- [Derived] Liu F, Zhang J, Zhu Y, Su L, Li Y, He L, Yu L, Peng Z. Acetate Ringer's solution versus 0.9% saline for septic patients: study protocol for a multi-center parallel controlled trial. Trials. 2021 Jan 25;22(1):89. doi: 10.1186/s13063-020-05007-5. PMID 33494795